CLINICAL TRIAL: NCT00444405
Title: Surgical Treatment Comparison for Recurrent Lumbar Disc Herniation
Status: Withdrawn | Type: Observational
Why Stopped: PI left Health System
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Michelle McFarland, MPH, CHRC, Manager - Mercy Research, Mercy Research
Other Study IDs: SJCNS-01
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain; Recurrent Lumbar Disc Herniation
Keywords: lumbar; disc; herniation; discectomy; fusion; spine
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement; Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to compare patients who underwent decompression/discectomy with pedicle screw fusion to patients who received decompression/discectomy without fusion.

DETAILED DESCRIPTION:
Lumbar disc herniations are quite common and typically improve after surgical correction. However, some patients develop recurrent herniations at the same level. Controversy exists as to why reherniated discs occur. Moreover, existing research does not settle the issue of whether a second decompression/discectomy or a repeat decompression/discectomy with pedicle screw fusion is the more successful treatment. This study is designed to compare differences in patient-reported pain, physical function, and satisfaction between the two types of surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent lumbar disc herniation by MRI or CT with history of decompression at the same level in the past
* Recurrent symptomatic history (with or without back pain) with radicular leg pain that improved following the first surgery
* Male or female 18-75 years old
* Flexion and extension x-rays that demonstrate an absence of sponylolisthesis or spondylolisthesis with less than 3 mm of movement

Exclusion Criteria:

* Recurrence of disc herniation within 3 months of first decompression
* Multiple level herniated discs
* No history of lumbar back surgery except as in Inclusion criteria above
* Documented severe osteoporosis or osteopenia
* Symptoms of low back pain only
* Diabetes mellitus
* Patients with suspected or diagnosed psychological/psychiatric problems that could compromise the reliability of their results
* Lumbar spondylolisthesis on flexion/extension x-rays > 3 mm
* History of lumbar spine fractures (new or old)
* Any concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study
* Autoimmune diseases
* Age less than 18 or greater than 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with recurrent lumbar disc herniation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan M. Scarrow, MD, JD, Principal Investigator — St. John's Health System, Missouri